CLINICAL TRIAL: NCT04023864
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Platycodon Grandiflorus Extract(GCWB107) on Decrease of Body Fat
Brief Title: Efficacy and Safety of Platycodon Grandiflorus Extract(GCWB107) on Decrease of Body Fat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCWB-BF-PG
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Body Fat
Keywords: Platycodon Grandiflorus Extract; Body Fat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platycodon Grandiflorus Extract(GCWB107) group (Experimental): Once-daily, once a tablet, after meals (900 mg/day, 571 mg/day as a Platycodon Grandiflorus Extract(GCWB107))
  Interventions: Dietary Supplement: Platycodon Grandiflorus Extract(GCWB107)
- Placebo group (Placebo Comparator): Once-daily, once a tablet, after meals (900 mg/day, 0 mg/day as a Platycodon Grandiflorus Extract(GCWB107))
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Platycodon Grandiflorus Extract(GCWB107) — Once-daily, once a tablet, after meals, for 12 week
  Arms: Platycodon Grandiflorus Extract(GCWB107) group
Dietary Supplement: Placebo — Placebo for 12 week
  Arms: Placebo group

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Platycodon grandiflorus extract(GCWB107) on decrease of body fat.

DETAILED DESCRIPTION:
This study was a 12-week, randomized, double-blind, placebo-controlled human trial. 80 subjects were randomly divided into Platycodon grandiflorus extract(GCWB107) group and a placebo group. It is to evaluate the changes in the displayed evaluation items when taking Platycodon grandiflorus extract(GCWB107) extract once a day, in comparison with taking a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 19 and 65 years at the screening
* Participants who were BMI 25~29.9 kg/m^2
* Participants who have fully understood the information provided about the study voluntarily decided to participate and agreed to comply with precautions

Exclusion Criteria:

* Participants who decrease 10% more of weight within 3 months period to the screening examination
* Participants taking for products affecting body weight within 4 weeks before the screening examination(i.e., Improvement of body fat Healthy functional food, contraceptive, steroid drug treatment, female hormone drug treatment) (However, participation is possible after a 4-week withdrawal period prior to the first intake day)
* Participants who drink more than 14 units/week of alcohol intake
* Patients with a clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry system, musculoskeletal system, inflammatory and hematologic
* Patients with diabetics who are taking oral hypoglycemic agents and insulin (at the screening)
* Participants with a past history of gastrointestinal diseases (e.g., Crohn's disease) or gastrointestinal surgery (but, excluding simple cecal surgery and hernia surgery) that can affect the absorption of products of the human trial
* Participants who have a history of clinically significant hypersensitivity to balloon flower and saponin components
* Participants receiving antipsychotic medication within 2 months prior to the screening examination
* Participants who were doubtful about drug abuse
* Participants who have participated in other clinical trials within 3 months prior to the screening examination
* Participants who have SBP≥180 mmHg and DBP≥110 mmHg
* Menopause women
* Participants who show the following relevant results in a Laboratory test

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dl
* Women who are pregnant or breastfeeding
* Women who may become pregnant and have not used appropriate contraceptives
* Participants who the principal investigator judged inappropriate for the participant in this study because of a laboratory test result, etc

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes of body fat mass | 0 week and 12 week
  Body fat mass was measured in study baseline and 12 week.

SECONDARY OUTCOMES:
Changes of percent body fat | 0 week and 12 week
  Measurement is made using dual-energy X-ray absorptiometry (DEXA / Hologic Discovery, USA). Left-arm, right arm, left leg, right leg, trunk, total will be reported percent body fat in %.
Changes of fat free mass | 0 week and 12 week
  Measurement is made using dual-energy X-ray absorptiometry (DEXA / Hologic Discovery, USA). Left-arm, right arm, left leg, right leg, trunk, total will be reported fat free mass in g.
Changes of Anthropometric indicators | Screening, 0 week, and 12 week
  Anthropometric indicators(i.e., weight, body mass index, waist circumference, hip circumference, waist-hip ratio) were measured in study screening, 0 weeks, and 12 weeks.
Changes of indicator of lipid metabolism | 0 week and 12 week
  Indicators of lipid metabolism(i.e., Total cholesterol, Triglyceride, LDL-cholesterol, HDL-cholesterol) were measured in the study for 0 weeks and 12 weeks.
Changes of Obesity-related hormone index | 0 week and 12 week
  Obesity-related hormone indexes(i.e., Adiponectin, Leptin)were measured in the study for 0 weeks and 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea